CLINICAL TRIAL: NCT05370989
Title: Technology-Based Parent School Program: Randomized Controlled Trial
Brief Title: Technology-Based Parent School Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ebru Kilicarslan Toruner, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 310472
Record Dates: First submitted 2022-04-23; First posted 2022-05-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Growth and Development; Child Rearing; Early Childhood Caries
Keywords: Parent school; Child; Toddler; Growth and Development

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-Based Parent School Program. (Experimental): Technology-Based Parent School Program. This program, developing parents' self-efficacy and parenting skills in child care with the Parent School Program
  Interventions: Other: Technology-Based Parent School Program; Other: ongoing treatment
- Control group (Active Comparator): the control group will continue to receive routine check-ups.
  Interventions: Other: ongoing treatment

INTERVENTIONS:
Other: Technology-Based Parent School Program — The program will be continued for 10 weeks in the intervention group and will be included five web-based modules, five online group interactions after each module, and consultation throughout the program and the follow-up period.
  Arms: Technology-Based Parent School Program.
Other: ongoing treatment — Health service of the control group will ongoing.

SUMMARY:
Objective: The purpose of this study was to assess the efficacy of a technology-based parent school program designed for parents of toddlers to be improved their parenting abilities.

Design: A parallel group, randomized controlled trial. Method: The study will be conducted with parents whose children are between the ages of 18 and 24 months in a hospital's well-child outpatient clinic in Turkey. The study data will be analyzed using the Parent and Child Descriptive Data Form, the Parent Skill List, Toddler Skill List, and the Turkish Version of Self-Efficacy for Parenting Tasks Index-Toddler Scale. The program will be continued for 10 weeks in the intervention group and will be included five web-based modules, five online group interactions after each module, and consultation throughout the program and the follow-up period. The modules will be included topics such as the child's physical growth, cognitive and linguistic development, and social-emotional development. The modules will be supported by videos and messages. This study will be based on Meleis' Transition Theory.

Hypothesis:

H0-1: There is no difference in self-efficacy total scores of parents between intervention and control group.

H0-2: There is no difference in parenting skill list total scores between intervention and control group.

H0-3: There is no difference in the skill list total scores of toddlers according to the parents between intervention and control group.

H1-1: There is a difference in self-efficacy total scores of parents between intervention and control group.

H1-2: There is a difference in parenting skill list total scores between intervention and control group.

H1-3: There is a difference in the skill list total scores of toddlers according to the parents between intervention and control group.

ELIGIBILITY:
Inclusion Criteria:

* to have given birth when you were 18 years and older
* to be parents whose children are between the ages of 16 and 21 months
* For the first time, having a child
* to be have internet access and smartphone or computer
* to agree to participate in the study

Exclusion Criteria:

* Parents who have a congenital defect, a chronic illness, or a mental disorder that their child has
* Prematurely born children
* Mothers who have been in their adolescents

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Parent Skill List | Change in parent skill level after 3 months
  The form was created by the researchers by scanning the literature. Contains 25 items. For their children's physical, cognitive-language, and social-emotional development, the form includes skills that parents can do, cannot do, or are hesitant to do. Parents will receive a minimum of 0 and a maximum of 50 points.
Toddler Skill List | Toddler skill level 3 months after the beginning of the program.
  The form was created by the researchers by scanning the literature. Contains 15 items. The form will evaluate what skills they have and what they will be unable to do for the physical, cognitive-language, and social-emotional development of toddlers. Toddler will receive a minimum of 0 and a maximum of 30 points.
the Turkish Version of Self-Efficacy for Parenting Tasks Index-Toddler Scale | Change in parent self-efficacy compliance from baseline at 3 months.
  The scale consists of 51 items to measure the self-efficacy of parents of children aged 1-3. The 5-point Likert-type scale is scored as 5: Totally Agree, 4: Agree, 3: Undecided, 2: Disagree, and 1: Strongly Disagree for positive items. Some of the items are scored reverse. The total score ranges from 51 to 255, with increasing scores indicating a high level of self-efficacy.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cirlak A, Kilicarslan E. Technology-based parent school: A randomized controlled trial. Public Health Nurs. 2024 Sep-Oct;41(5):1188-1198. doi: 10.1111/phn.13371. Epub 2024 Jul 16. PMID 39010780